CLINICAL TRIAL: NCT01588496
Title: 2-part, Phase 2/3 Study to Assess the Safety, Tolerability and Efficacy of AMG 145 in Subjects With Homozygous Familial Hypercholesterolemia. Part A - Open-label, Single-arm, Multicenter Pilot Study to Evaluate Safety, Tolerability and Efficacy of AMG 145 in Subjects With Homozygous Familial Hypercholesterolemia. Part B - Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate Safety, Tolerability and Efficacy of AMG 145 in Subjects With Homozygous Familial Hypercholesterolemia
Brief Title: Trial Evaluating PCSK9 Antibody in Subjects With LDL Receptor Abnormalities
Acronym: TESLA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110233; 2011-005399-40 (EudraCT Number)
Record Dates: First submitted 2012-02-27; First posted 2012-05-01 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: hypercholesterolemia; familial hypercholesterolemia; homozygous familial hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part A: Evolocumab (Experimental): Participants received open-label evolocumab 420 mg subcutaneously once a month for 12 weeks.
  Interventions: Biological: Evolocumab
- Part B: Evolocumab (Experimental): Participants received double-blind evolocumab 420 mg subcutaneously once a month for 12 weeks.
  Interventions: Biological: Evolocumab
- Part B: Placebo (Placebo Comparator): Participants received double-blind placebo subcutaneously once a month for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Part A: Evolocumab; Part B: Evolocumab
Drug: Placebo — Administered by subcutaneous injection
  Arms: Part B: Placebo

SUMMARY:
A study to determine the safety, tolerability, and efficacy of evolocumab (AMG 145) in patients with homozygous familial hypercholesterolemia (HoFH).

DETAILED DESCRIPTION:
Study Masking:

Part A: Open Label Part B: Double Blind

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 12 to ≤ 80 years of age
* Diagnosis of homozygous familial hypercholesterolemia
* Stable lipid-lowering therapies for at least 4 weeks
* LDL cholesterol ≥ 130 mg/dl (3.4 mmol/L)
* Triglyceride ≤ 400 mg/dL (4.5 mmol/L)
* Bodyweight of ≥ 40 kg at screening.

Exclusion Criteria:

* LDL or plasma apheresis within 8 weeks prior to randomization
* New York Heart Association (NYHA) class III or IV or last known left ventricular ejection fraction < 30%
* Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke within 3 months of randomization
* Planned cardiac surgery or revascularization
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-04-05 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2014-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (21):
- United States (2):
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
- Belgium (2):
  - Research Site, Brussels
  - Research Site, La Louvière
- Canada (2):
  - Research Site, London, Ontario
  - Research Site, Chicoutimi, Quebec
- Czechia (3):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Uherské Hradiště
- France (2):
  - Research Site, Dijon
  - Research Site, Paris
- Research Site, New Territories, Hong Kong
- Research Site, Pisa, Italy
- Research Site, Beirut, Lebanon
- Research Site, Amsterdam, Netherlands
- Research Site, Christchurch, New Zealand
- South Africa (2):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Observatory, Western Cape
- Spain (3):
  - Research Site, Córdoba, Andalusia
  - Research Site, Lugo, Galicia
  - Research Site, Madrid

REFERENCES:
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Derived] Raal FJ, Honarpour N, Blom DJ, Hovingh GK, Xu F, Scott R, Wasserman SM, Stein EA; TESLA Investigators. Inhibition of PCSK9 with evolocumab in homozygous familial hypercholesterolaemia (TESLA Part B): a randomised, double-blind, placebo-controlled trial. Lancet. 2015 Jan 24;385(9965):341-50. doi: 10.1016/S0140-6736(14)61374-X. Epub 2014 Oct 1. PMID 25282520
- [Derived] Stein EA, Honarpour N, Wasserman SM, Xu F, Scott R, Raal FJ. Effect of the proprotein convertase subtilisin/kexin 9 monoclonal antibody, AMG 145, in homozygous familial hypercholesterolemia. Circulation. 2013 Nov 5;128(19):2113-20. doi: 10.1161/CIRCULATIONAHA.113.004678. Epub 2013 Sep 6. PMID 24014831
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female adults and adolescents ages ≥ 12 to ≤ 65 years (≥ 12 to ≤ 80 years in Part B) with a diagnosis of homozygous familial hypercholesterolemia (HoFH) were eligible for this study. The first participant enrolled on 05 April 2012 and the last participant enrolled on 08 November 2013.
Pre-assignment Details: Part A was an open-label, single-arm, multicenter pilot study. Part B was a double-blind, randomized, placebo-controlled, multicenter study with expanded enrollment. In Part B participants were randomized in a 1:2 allocation stratified on the basis of screening low-density lipoprotein cholesterol (LDL-C) (< 420 mg/dL vs ≥ 420 mg/dL).
Groups:
- Part A: Evolocumab: Participants received open-label evolocumab 420 mg subcutaneously (SC) once a month (QM) for 12 weeks.
Period: Overall Study
Arm/Group | Part A: Evolocumab | Part B: Placebo | Part B: Evolocumab
Started | 8 | 17 | 33
Received Treatment | 8 | 16 | 33
Completed | 8 | 16 | 33
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Evolocumab | Part B: Placebo | Part B: Evolocumab | Total
Number analyzed (Participants) | 8 | 17 | 33 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (12.4) | 32.8 (13.7) | 30.3 (12.4) | 31.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 16 | 26
  Male | 6 | 9 | 17 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Black or African American | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 8 | 16 | 29 | 53
  Other | 0 | 0 | 3 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 17 | 32 | 57
Stratification Factor: Low-Density Lipoprotein Cholesterol (LDL-C) Level [Number; unit: participants] — Participants in Part A were not stratified based on LDL-C level.
  participants
    < 420 mg/dL | 0 | 11 | 21 | 32
    ≥ 420 mg/dL | 0 | 6 | 12 | 18
    Missing | 8 | 0 | 0 | 8
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] — LDL-C was quantified using the ultracentrifugation method. Data are provided for the full analysis set (all enrolled participants who received at least 1 dose of evolocumab (Part A) or all randomized participants who received at least 1 dose of investigational product (Part B).
  mg/dL
    Part A | 441.7 (113.3) | NA (NA) — Not applicable for Part B participants | NA (NA) — Not applicable for Part B participants | 441.7 (113.3)
    Part B | NA (NA) — Not applicable for Part A participants | 335.8 (146.0) | 356.0 (134.5) | 349.4 (137.2)
Non-High-Density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL
    Part A | 470.6 (117.8) | NA (NA) — Not applicable for Part B participants | NA (NA) — Not applicable for Part B participants | 470.6 (117.8)
    Part B | NA (NA) — Not applicable for Part A participants | 358.9 (149.1) | 374.9 (136.9) | 369.7 (139.6)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL
    Part A | 269.1 (53.0) | NA (NA) — Not applicable for Part B participants | NA (NA) — Not applicable for Part B participants | 269.1 (53.0)
    Part B | NA (NA) — Not applicable for Part A participants | 208.6 (79.5) | 208.3 (68.4) | 208.4 (71.4)
Total Cholesterol/HDL-C Ratio [Mean (Standard Deviation); unit: ratio] — Data are provided for the full analysis set
  ratio
    Part A | 15.988 (5.107) | NA (NA) — Not applicable for Part B participants | NA (NA) — Not applicable for Part B participants | 15.988 (5.107)
    Part B | NA (NA) — Not applicable for Part A participants | 12.101 (6.619) | 11.972 (6.387) | 12.014 (6.395)
Apolipoprotein B/Apolipoprotein A1 Ratio [Mean (Standard Deviation); unit: ratio] — Data are provided for the full analysis set
  ratio
    Part A | 2.800 (0.729) | NA (NA) — Not applicable for Part B participants | NA (NA) — Not applicable for Part B participants | 2.800 (0.729)
    Part B | NA (NA) — Not applicable for Part A participants | 2.053 (0.967) | 2.098 (1.046) | 2.084 (1.011)
Lipoprotein(a) Concentration [Median (Inter-Quartile Range); unit: nmol/L]
  Part A | 246.5 [61.5 to 276] | NA [NA to NA] — Not applicable for Part B participants | NA [NA to NA] — Not applicable for Part B participants | 246.5 [61.5 to 276]
  Part B | NA [NA to NA] — Not applicable for Part A participants | 127.5 [79.5 to 200.5] | 76.0 [25.5 to 145.0] | 100.5 [31.0 to 146.0]
Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Concentration [Mean (Standard Deviation); unit: ng/mL] — Data are provided for the full analysis set
  ng/mL
    Part A | 598.6 (121.1) | NA (NA) — Not applicable for Part B participants | NA (NA) — Not applicable for Part B participants | 598.6 (121.1)
    Part B | NA (NA) — Not applicable for Part A participants | 674.2 (180.0) | 640.3 (207.5) | 651.4 (197.7)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: LDL-C was quantified using the ultracentrifugation method.
Time Frame: Baseline and Week 12
Population: Part A full analysis set (all enrolled participants who received at least 1 dose of evolocumab)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part A: Evolocumab
Number analyzed (Participants) | 8
percent change | -16.5 (6.7)

2. Secondary Outcome: Part A: Change From Baseline in LDL-C at Week 12
Description: LDL-C was quantified using the ultracentrifugation method.
Time Frame: Baseline and Week 12
Population: Part A full analysis set
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Part A: Evolocumab
Number analyzed (Participants) | 8
mg/dL | -70.6 (32.3)

3. Secondary Outcome: Part A: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Part A full analysis set
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part A: Evolocumab
Number analyzed (Participants) | 8
percent change | -16.6 (6.5)

4. Secondary Outcome: Part A: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and Week 12
Population: Part A full analysis set
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part A: Evolocumab
Number analyzed (Participants) | 8
percent change | -14.9 (5.0)

5. Secondary Outcome: Part A: Percent Change From Baseline in the Total Cholesterol/HDL-C Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Part A full analysis set
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part A: Evolocumab
Number analyzed (Participants) | 8
percent change | -18.319 (6.058)

6. Secondary Outcome: Part A: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Part A full analysis set
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part A: Evolocumab
Number analyzed (Participants) | 8
percent change | -15.65 (4.690)

7. Secondary Outcome: Part A: Percentage of Participants With 15% or Greater Reduction in LDL-C From Baseline at Week 12
Description: LDL-C was quantified using the ultracentrifugation method.
Time Frame: Baseline and Week 12
Population: Part A full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Evolocumab
Number analyzed (Participants) | 8
percentage of participants | 50.0

8. Secondary Outcome: Part A: Change From Baseline in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) at Week 12
Time Frame: Baseline and Week 12
Population: Part A full analysis set
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Part A: Evolocumab
Number analyzed (Participants) | 8
ng/mL | -151.3 (81.7)

9. Secondary Outcome: Part B: Percent Change From Baseline in LDL-C at the Mean of Weeks 6 and 12
Description: LDL-C was quantified using the ultracentrifugation method.
Time Frame: Baseline and Weeks 6 and 12
Population: Part B full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part B: Placebo | Part B: Evolocumab
Number analyzed (Participants) | 16 | 33
percent change | 4.22 (4.56) | -25.56 (3.28)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Model includes treatment group, baseline LDL-C level (< 420 vs ≥ 420 mg/dL), scheduled visit and the interaction of treatment with scheduled visit; LS Mean Treatment Difference = -29.78, 95% CI 2-sided [-40.94 to -18.62], Standard Error of Mean 5.54 — Placebo is the reference

10. Secondary Outcome: Part B: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and Week 12
Population: Part B full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part B: Placebo | Part B: Evolocumab
Number analyzed (Participants) | 16 | 33
percent change | 3.97 (4.74) | -19.17 (3.46)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 9, analysis 1]; LS Mean Treatment Difference = -23.14, 95% CI 2-sided [-34.83 to -11.45], Standard Error of Mean 5.81 — Placebo is the reference

11. Secondary Outcome: Part B: Percent Change From Baseline in Apolipoprotein B at the Mean of Weeks 6 and 12
Time Frame: Baseline and Weeks 6 and 12
Population: Part B full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part B: Placebo | Part B: Evolocumab
Number analyzed (Participants) | 16 | 33
percent change | 2.65 (4.42) | -20.24 (3.18)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 9, analysis 1]; LS Mean Treatment Difference = -22.89, 95% CI 2-sided [-33.72 to -12.05], Standard Error of Mean 5.38 — Placebo is the reference

12. Secondary Outcome: Part B: Percent Change From Baseline in Lipoprotein (a) at Week 12
Time Frame: Baseline and Week 12
Population: Part B full anlaysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part B: Placebo | Part B: Evolocumab
Number analyzed (Participants) | 16 | 33
percent change | 2.43 (5.49) | -9.40 (4.07)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: Evolocumab; Test type: Superiority or Other; p = 0.088, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 9, analysis 1]; LS Mean Treatment Difference = -11.83, 95% CI 2-sided [-25.48 to 1.82], Standard Error of Mean 6.77 — Placebo is the reference

13. Secondary Outcome: Part B: Percent Change From Baseline in Lipoprotein (a) at the Mean of Weeks 6 and 12
Time Frame: Baseline and Weeks 6 and 12
Population: Part B full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part B: Placebo | Part B: Evolocumab
Number analyzed (Participants) | 16 | 33
percent change | -1.43 (4.78) | -12.71 (3.53)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: Evolocumab; Test type: Superiority or Other; p = 0.088, Repeated measures linear effects — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 9, analysis 1]; LS Mean Treatment Difference = -11.27, 95% CI 2-sided [-23.11 to 0.56], Standard Error of Mean 5.86 — Placebo is the reference

14. Primary Outcome: Part B: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: LDL-C was quantified using the ultracentrifugation method.
Time Frame: Baseline and Week 12
Population: Part B full analysis set (all enrolled participants who received at least 1 dose of investigational product)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part B: Placebo | Part B: Evolocumab
Number analyzed (Participants) | 16 | 33
percent change | 7.88 (5.26) | -23.05 (3.78)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: Evolocumab; LDL-C lowering was analyzed by comparing evolocumab and placebo. Statistical analysis was 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 9, analysis 1]; LS Mean Treatment Difference = -30.93, 95% CI 2-sided [-43.86 to -18.00], Standard Error of Mean 6.42 — Placebo is the reference

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
  MedDRA 16.0 was used to code adverse events in Part A; MedDRA 16.1 was used to code adverse events in Part B.
Groups:
- Part A: OL Evolocumab: Participants received open-label (OL) evolocumab 420 mg subcutaneously once a month for 12 weeks.
- Part B: DB Placebo: Participants received double-blind (DB) placebo subcutaneously once a month for 12 weeks.
- Part B: DB Evolocumab: Participants received double-blind evolocumab 420 mg subcutaneously once a month for 12 weeks.
Arm/Group | Part A: OL Evolocumab | Part B: DB Placebo | Part B: DB Evolocumab
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/16 | 0/33
Other Adverse Events (participants affected / at risk) | 4/8 | 10/16 | 11/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: OL Evolocumab (N=8) | Part B: DB Placebo (N=16) | Part B: DB Evolocumab (N=33)
Palpitations (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Chest pain (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Medical device site reaction (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.